CLINICAL TRIAL: NCT05707286
Title: Pilot Study to Determine Pro-Inflammatory Cytokine Kinetics During Immune Checkpoint Inhibitor Therapy
Acronym: ICI-PICK
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Tyler Andrew Shugg, Assistant Research Professor, Indiana University
Other Study IDs: CPHR-IIR-CYTOKINE; K23GM147805 (NIH)
Record Dates: First submitted 2023-01-20; First posted 2023-01-31 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Melanoma; Gastrointestinal Neoplasms; Genitourinary Cancer; Thoracic Cancer; Sarcoma
Keywords: Checkpoint inhibitor; cytokines
MeSH Terms: conditions — Melanoma; Gastrointestinal Neoplasms; Urogenital Neoplasms; Sarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — This study is observational in nature and will involve no medical interventions outside of collecting 5-7 blood samples at 5-7 separate study visits.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This research aims to identify clinical strategies to manage adverse events during immune checkpoint inhibitor therapy by (1) determining the impact of checkpoint inhibitors on metabolism through major CYP enzymes and (2) identifying associations between pro-inflammatory cytokine concentrations and negative clinical outcomes during checkpoint inhibitor therapy.

DETAILED DESCRIPTION:
The long-term goal of this research is to identify clinical strategies to manage adverse events during checkpoint inhibitor therapy. The research aims of the current project are (1) to determine the impact of checkpoint inhibitor therapy on the metabolism of CYP probe drugs and the risk for adverse events with CYP substrate drugs commonly prescribed to cancer patients and (2) to identify associations between pro-inflammatory cytokine concentrations and CYP probe drug metabolism before and during checkpoint inhibitor therapy. To investigate these aims, we plan to conduct a two-phase crossover clinical drug interaction study in which a cocktail containing probe drugs for six CYP enzymes (CYP1A2, CYP2B6, CYP2C9, CYP2C19, CYP2D6, and CYP3A) is administered to subjects before and after they initiate checkpoint inhibitor therapy. However, the kinetics of changes in pro-inflammatory cytokines during checkpoint inhibitor therapy are not well established, and this knowledge is critical to inform timing of the on-treatment phase of the clinical drug interaction study. Accordingly, this pilot study will investigate when blood concentrations of pro-inflammatory cytokines peak after initiation of checkpoint inhibitor therapy. Blood cytokine concentrations will be assayed at baseline, ~7 and ~14 days following the first checkpoint inhibitor cycle (± 2 days surrounding each timepoint), and at cycles 2, 3, and 4 based on the strongest current in vitro (7-14 days) and clinical evidence (21-42 days). In addition to plasma concentrations of pro-inflammatory cytokines, the study will also assay plasma concentrations of immune checkpoint inhibitors, co-administered CYP substrates, and perform genetic sequencing to assess associations between these variables and clinical outcomes, including the development of immune-related adverse events, the potential for drug-drug interactions with CYP substrates, and checkpoint inhibitor treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old at the time of informed consent
2. Diagnosed with non-small cell lung cancer (NSCLC) OR melanoma AND initiating therapy with single agent or combination therapy that includes an immune checkpoint inhibitor, (e.g., atezolizumab, cemiplimab, durvalumab, ipilimumab, nivolumab, pembrolizumab)
3. Ability to provide written informed consent and HIPAA authorization

Exclusion Criteria:

1. Diagnosis or past medical history of autoimmune disorder, including systemic lupus erythematosus, Crohn's disease, Sjogren's syndrome, multiple sclerosis, type 1 diabetes mellitus, Behcet's disease, and ankylosing spondylitis
2. Current infection requiring medical treatment (note: if a prospective subject's infection resolves, they can be re-screened for trial inclusion)
3. Concomitant treatment with systemic immunosuppressant drugs (see Table A1 in appendix for complete list)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with solid cancers and initiating therapy with an immune checkpoint inhibitor
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2023-09-07 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Increases in pro-inflammatory cytokines | From baseline (day -30) up to cycle 4 (day 126)
  Determine the time course of increases in pro-inflammatory cytokines during treatment with immune checkpoint inhibitor regimens, via plasma cytokine concentrations present in blood samples.
Populations of activated T cells | From baseline (day -30) up to cycle 4 (day 126)

SECONDARY OUTCOMES:
Increases in other cytokines | From baseline (day -30) up to cycle 4 (day 126)
  Determine the time course of increases in other cytokines during treatment with immune checkpoint inhibitor regimens, including anti-inflammatory cytokines (e.g., IL-10, TGF-β) present in blood samples.
Plasma concentrations of immune checkpoint inhibitors | From baseline (day -30) up to cycle 4 (day 126)
  Assess on-treatment concentrations of immune checkpoint inhibitors
Plasma concentrations of co-administered CYP substrate medications | From baseline (day -30) up to cycle 4 (day 126)
  Assess baseline and on-treatment concentrations of co-administered CYP substrate medications
The development of immune-related adverse events | From baseline (day -30) up to cycle 4 (day 126)
  Immune-related adverse events will be assessed via patient survey at all study visits
The development of adverse drug events attributable to co-administered CYP substrate medications | From baseline (day -30) up to cycle 4 (day 126)
  Adverse drug events attributable to co-administered CYP substrate medications will be assessed via patient survey at all study visits
Checkpoint inhibitor treatment response | From treatment initiation (day 0) until the time of the treatment response event or the end of the study evaluation period (maximum of 2 years from the date of treatment initiation).
  Checkpoint inhibitor treatment response will be collected retrospectively from the electronic health record

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Shugg, PharmD, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana, United States